CLINICAL TRIAL: NCT01138657
Title: A Multicenter Study of the Efficacy and Safety of the Human Anti-TNF Monoclonal Antibody Adalimumab as Maintenance Therapy in Subjects Requiring High Dose Corticosteroids for Active Non-infectious Intermediate Uveitis, Posterior Uveitis, or Panuveitis - Including a Sub-study in Japanese Patients
Brief Title: Efficacy and Safety of Adalimumab in Patients With Active Uveitis
Acronym: VISUAL l
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-877; 2009-016095-68 (EudraCT Number)
Record Dates: First submitted 2010-05-14; First posted 2010-06-07 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Uveitis
Keywords: inflammation of uvea
MeSH Terms: conditions — Uveitis | interventions — Adalimumab; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adalimumab (Experimental): Participants received adalimumab 80 mg subcutaneous loading dose at Baseline followed by 40 mg doses every other week (eow) starting at Week 1 for a maximum of 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 60 mg/day at study entry followed by a protocol-defined mandatory taper until Week 15.
  Interventions: Biological: Adalimumab; Drug: Prednisone
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection at Baseline followed by eow dosing starting at Week 1 for up to 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 60 mg/day at study entry followed by a protocol-defined mandatory taper until Week 15.
  Interventions: Drug: Prednisone; Drug: Placebo

INTERVENTIONS:
Biological: Adalimumab — Administered subcutaneously as an 80 mg loading dose (2 syringes) at Baseline followed by a 40 mg dose eow starting at Week 1.
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab
Drug: Prednisone — Administered orally, 60 mg/day at study entry followed by a protocol-defined mandatory taper schedule in which all participants continuing in the study were to discontinue prednisone no later than Week 15.
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
A study comparing the safety and efficacy of adalimumab compared with placebo in patients with active uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject is diagnosed with non-infectious intermediate-, posterior-, or panuveitis.
* Subject must have active disease at the Baseline visit as defined by the presence of at least 1 of the following parameters in at least one eye despite at least 2 weeks of maintenance therapy with oral prednisone ≥ 10 mg/day to ≤ 60 mg/day (or oral corticosteroid equivalent):

  * Active, inflammatory, chorioretinal and/or inflammatory retinal vascular lesion
  * ≥ 2+ anterior chamber cells (Standardization of Uveitis Nomenclature [SUN] criteria)
  * ≥ 2+ vitreous haze (National Eye Institute [NEI]/SUN criteria)
* Subject is on oral prednisone ≥ 10 mg/day to ≤ 60 mg/day (or oral corticosteroid equivalent) for at least 2 weeks prior to Screening and remains on the same dose from Screening to Baseline visit.
* Subject with documented prior adequate response to oral corticosteroids (equivalent of oral prednisone up to 1 mg/kg/day).
* Subjects who do not have previous, active or latent tuberculosis (TB). Only one TB test is required to allow the subject in the study. Subjects with either negative purified protein derivative (PPD) (< 5 mm of induration) or negative QuantiFERON®-TB Gold test (or interferon-gamma release assay (IGRA) equivalent) are eligible. Subjects with a repeat indeterminate QuantiFERON®-TB Gold test (or IGRA equivalent) result are not eligible. Note, that only one TB screening test is allowed and required. A repeat QuantiFERON® TB Gold test (or IGRA equivalent) is not permitted if the PPD skin test is positive. The TB screening tests are diagnostic tests. In the event of a negative TB screening test, the results are to be interpreted in the context of the patient's epidemiology, history, exam findings, etc. and it is the responsibility of the investigator to determine if a patient has previous, active or latent tuberculosis or not. Under no circumstances can a patient with a positive PPD result or positive QuantiFERON®-TB Gold test (or IGRA equivalent) enter the study.

Exclusion Criteria:

* Subject with isolated anterior uveitis.
* Subject with prior inadequate response to high-dose oral corticosteroids
* Subject with confirmed or suspected infectious uveitis, including but not limited to infectious uveitis due to TB, cytomegalovirus (CMV), Human T-Lymphotropic Virus Type 1 (HTLV-1), Whipple's disease, Herpes Zoster virus (HZV), Lyme disease, toxoplasmosis and herpes simplex virus (HSV).
* Subject with serpiginous choroidopathy.
* Subject with corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the trial.
* Subject with intraocular pressure of ≥ 25 mmHg and on ≥ 2 glaucoma medications or evidence of glaucomatous optic nerve injury.
* Subject with Best Corrected Visual Acuity (BCVA) less than 20 letters (Early Treatment Diabetic Retinopathy Study) in at least one eye at the Baseline Visit.
* Subject with intermediate uveitis or panuveitis that has signs of intermediate uveitis (e.g.presence or history of snowbanking or snowballs) and symptoms and/or magnetic resonance imaging (MRI) findings suggestive of a demyelinating disease such as multiple sclerosis. All subjects with intermediate uveitis or panuveitis that have signs of intermediate uveitis (e.g., presence or history of snowbanking or snowballs) must have had a brain MRI within 90 days prior to the Baseline Visit.
* Subject has previous exposure to anti-tumor necrosis factor (TNF) therapy or any biologic therapy (except intravitreal anti-vascular endothelial growth factor [VEGF] therapy) with a potential therapeutic impact on non-infectious uveitis.
* If entering the study on 1 concomitant immunosuppressive therapy, dose has been increased within the last 28 days prior to Baseline visit or is not within the following allowable doses at the Baseline visit:

  * Methotrexate (MTX) ≤ 25 mg per week
  * Cyclosporine ≤ 4 mg/kg per day
  * Mycophenolate mofetil ≤ 2 grams per day or an equivalent drug to mycophenolate mofetil (e.g. mycophenolic acid) at an equivalent dose approved by the Medical Monitor.
  * Azathioprine ≤ 175 mg per day
  * Tacrolimus (oral formulation) ≤ 8 mg per day
* Subject has received Retisert® (glucocorticosteroids implant) within 3 years prior to the Baseline visit or that has had complications related to the device. Subject has had Retisert® (glucocorticosteroids implant) removed within 90 days prior to the Baseline visit or has had complications related to the removal of the device.
* Subject has received intraocular or periocular corticosteroids within 30 days prior to Baseline visit.
* Subject with proliferative or severe non-proliferative diabetic retinopathy or clinically significant macular edema due to diabetic retinopathy.
* Subject with neovascular/wet age-related macular degeneration
* Subject with abnormality of vitreo-retinal interface (i.e., vitreomacular traction, epiretinal membranes, etc.) with the potential for macular structural damage independent of the inflammatory process.
* Subject with severe vitreous haze that precludes visualization of the fundus at the Baseline visit.
* Subject has received Ozurdex® (dexamethasone implant) within 6 months prior to the Baseline visit.
* Subject has received intravitreal anti-VEGF therapy within 45 days of the Baseline visit for Lucentis® (ranibizumab) or Avastin® (bevacizumab) or within 60 days of the Baseline visit for anti-VEGF Trap (aflibercept).
* Subject has received intravitreal methotrexate within 90 days prior to the Baseline visit
* Subject on systemic carbonic anhydrase inhibitor within 1 week prior to Screening visit.
* Subject with macular edema as the only sign of uveitis.
* Subject with a history of scleritis.
* Subject with intolerance to high-dose oral corticosteroids (equivalent of oral prednisone 1 mg/kg/day or 60 to 80 mg/day).
* Subject on cyclophosphamide within 30 days prior to the Baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2010-08; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Payne, PhD, Study Director — AbbVie

REFERENCES:
- [Result] Jaffe GJ, Dick AD, Brezin AP, Nguyen QD, Thorne JE, Kestelyn P, Barisani-Asenbauer T, Franco P, Heiligenhaus A, Scales D, Chu DS, Camez A, Kwatra NV, Song AP, Kron M, Tari S, Suhler EB. Adalimumab in Patients with Active Noninfectious Uveitis. N Engl J Med. 2016 Sep 8;375(10):932-43. doi: 10.1056/NEJMoa1509852. PMID 27602665
- [Derived] Sheppard J, Joshi A, Betts KA, Hudgens S, Tari S, Chen N, Skup M, Dick AD. Effect of Adalimumab on Visual Functioning in Patients With Noninfectious Intermediate Uveitis, Posterior Uveitis, and Panuveitis in the VISUAL-1 and VISUAL-2 Trials. JAMA Ophthalmol. 2017 Jun 1;135(6):511-518. doi: 10.1001/jamaophthalmol.2017.0603. PMID 28426849
- [Derived] Grewal DS, O'Sullivan ML, Kron M, Jaffe GJ. Association of Disorganization of Retinal Inner Layers With Visual Acuity In Eyes With Uveitic Cystoid Macular Edema. Am J Ophthalmol. 2017 May;177:116-125. doi: 10.1016/j.ajo.2017.02.017. Epub 2017 Feb 22. PMID 28237411
- See also: This clinical study may be evaluating a usage that is not currently FDA-approved. Please see US Prescribing Information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study includes a Japan sub-study. 239 participants with active non-infectious intermediate uveitis, posterior uveitis, or panuveitis were randomized worldwide, including 223 participants at 67 sites in Australia, Europe, Israel, Latin America, and North America (Main Study), and 16 participants randomized at 7 sites in Japan (Japan sub-study).
Pre-assignment Details: Participants were randomized in a 1:1 ratio double-masked fashion stratified by baseline immunosuppressant usage. Participants recruited in the Japan sub-study were randomized in a separate stratum with no stratification by baseline immunosuppressant usage.
  Study completion was defined as meeting treatment failure or reaching study Week 80.
Groups:
- Placebo: Participants received placebo subcutaneous injection at Baseline followed by every other week (eow) dosing starting at Week 1 for up to 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 60 mg/day at study entry followed by a protocol-defined mandatory taper until Week 15.
- Adalimumab: Participants received adalimumab 80 mg subcutaneous loading dose at Baseline followed by 40 mg doses eow starting at Week 1 for a maximum of 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 60 mg/day at study entry followed by a protocol-defined mandatory taper until Week 15.
Period: Overall Study
Arm/Group | Placebo | Adalimumab
Started | 120 | 119
Enrolled in Main Study | 112 | 111
Enrolled in Japan Sub-study | 8 | 8
Completed | 112 | 101
Not Completed | 8 | 18
Not completed — Adverse Event | 3 | 10
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 0 | 3
Not completed — Miscellaneous Reasons | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab | Total
Number analyzed (Participants) | 120 | 119 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.19 (14.331) | 43.46 (15.458) | 43.33 (14.872)
Age, Customized [Number; unit: participants]
  < 40 years | 56 | 47 | 103
  40 - 64 years | 54 | 56 | 110
  ≥ 65 years | 10 | 16 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 66 | 139
  Male | 47 | 53 | 100
Race/Ethnicity, Customized [Number; unit: participants]
  White | 91 | 89 | 180
  Black | 12 | 11 | 23
  Asian | 10 | 12 | 22
  American Indian/Alaskan Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 5 | 6 | 11
  Multi Race | 1 | 1 | 2
Type of Uveitis [Number; unit: participants]
  Intermediate | 24 | 25 | 49
  Posterior | 38 | 38 | 76
  Panuveitis | 58 | 56 | 114
Diagnosis [Number; unit: participants]
  Idiopathic | 50 | 40 | 90
  Birdshot Choroidopathy | 21 | 24 | 45
  Multifocal Choroiditis And Panuveitis | 5 | 8 | 13
  Vogt Koyanagi Harada | 14 | 12 | 26
  Sarcoid | 12 | 12 | 24
  Behcet's | 4 | 14 | 18
  Other | 14 | 9 | 23
Eye Affected [Number; unit: participants]
  Left | 5 | 6 | 11
  Right | 4 | 7 | 11
  Both | 111 | 106 | 217
Duration of Uveitis [Mean (Standard Deviation); unit: months] | 58.56 (85.308) | 41.18 (53.530) | 49.90 (71.660)

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure on or After Week 6
Description: Time to treatment failure was analyzed using Kaplan-Meier methods. Treatment failures on or after Week 6 were counted as events. Dropouts for reasons other than treatment failure at any time during the study were censored at the dropout date. To be considered a treatment failure, ≥ 1 of these criteria had to be present in at least 1 eye:
  * New active, inflammatory chorioretinal or retinal vascular lesions relative to Baseline
  * Inability to achieve ≤ 0.5+ at Week 6 or a 2-step increase relative to best state achieved at all visits after Week 6 in anterior chamber cell grade or vitreous haze grade
  * Worsening of best corrected visual acuity by ≥ 15 letters relative to best state achieved.
  Per protocol, the primary analysis was performed in the Main Study population which included all randomized participants recruited outside Japan; for completeness results are also reported below for the Integrated dataset which includes participants recruited in Japan.
Time Frame: From Baseline until end of study (up to 80 weeks)
Population: The intent-to-treat (ITT) population which included all randomized participants; 6 participants at 2 sites were excluded from the ITT due to incomplete efficacy source data and compliance issues.
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- Main Study: Placebo: Participants, excluding those enrolled in the Japan sub-study, received placebo subcutaneous injection at Baseline followed by eow dosing starting at Week 1 for up to 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 60 mg/day at study entry followed by a protocol-defined mandatory taper until Week 15.
- Main Study: Adalimumab: Participants, excluding those enrolled in the Japan sub-study, received adalimumab 80 mg subcutaneous loading dose at Baseline followed by 40 mg doses every other week (eow) starting at Week 1 for a maximum of 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 60 mg/day at study entry followed by a protocol-defined mandatory taper until Week 15.
- Integrated Study (Main + Japan Sub-study): Placebo: Participants, including those enrolled in the Main Study and the Japan Sub-study, received placebo subcutaneous injection at Baseline followed by eow dosing starting at Week 1 for up to 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 60 mg/day at study entry followed by a protocol-defined mandatory taper until Week 15.
- Integrated Study (Main + Japan Sub-study): Adalimumab: Participants, including those enrolled in the Main Study and the Japan Sub-study, received adalimumab 80 mg subcutaneous loading dose at Baseline followed by 40 mg doses every other week (eow) starting at Week 1 for a maximum of 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 60 mg/day at study entry followed by a protocol-defined mandatory taper until Week 15.
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 107 | 110 | 115 | 118
months | 3.0 [1.5 to 5.6] | 5.6 [3.0 to NA] — Not estimable due to the low number of events | 3.0 [1.5 to 5.6] | 4.8 [2.8 to NA] — Not estimable due to the low number of events
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; The primary analysis of the primary endpoint was performed on Main Study data, excluding the Japanese sub-study. The statistical test was performed at a 2-sided significance level of 0.05. The hazard ratio of adalimumab versus placebo was calculated using proportional hazards regression with treatment as factor; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.36 to 0.70]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; An additional analysis of the primary endpoint was performed using the Integrated Study data (Main Study + Japan sub-study). The statistical test was performed at a 2-sided significance level of 0.05. The hazard ratio of adalimumab versus placebo was calculated using proportional hazards regression with treatment and race (Japanese versus non-Japanese) as factors; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.40 to 0.76]

2. Secondary Outcome: Change in Anterior Chamber (AC) Cell Grade in Each Eye From Best State Achieved Prior to Week 6 to the Final/Early Termination Visit
Description: Slit lamp examinations were conducted at each visit to assess AC cell count. The number of AC cells observed within a 1 mm × 1 mm slit beam was used to determine the grade according to the Standardization of Uveitis Nomenclature (SUN) criteria:
  Grade 0 = < 1 cell;
  Grade 0.5+ = 1-5 cells;
  Grade 1+ = 6-15 cells;
  Grade 2+ = 16-25 cells;
  Grade 3+ = 26-50 cells;
  Grade 4+ = > 50 cells.
Time Frame: From Baseline to Week 6 and at the Final/Early Termination Visit (up to 80 weeks)
Population: Intent-to-treat population with values at both time points (best state achieved prior to Week 6 and at least 1 post-week 6 value); last observation carried forward (LOCF) imputation was used; participants with no values after Week 6 were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 102 | 101 | 110 | 109
units on a scale
  Left Eye | 0.59 (0.935) | 0.35 (0.763) | 0.56 (0.913) | 0.35 (0.744)
  Right Eye | 0.69 (1.067) | 0.36 (0.746) | 0.65 (1.039) | 0.36 (0.727)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; The statistical test for the ranked secondary variables was carried out in hierarchical order at the significance level of 5%; Test type: Superiority or Other; p = 0.011, ANOVA; ANOVA with treatment as factor adjusted for clustered observations (i.e., observations from each of the participant's eyes); Mean Difference = -0.29, 95% CI 2-sided [-0.51 to -0.07] — The mean difference between treatment groups with its 95% confidence interval is based on individual data from all eyes adjusted for correlated measurements within a subject in an analysis of variance (ANOVA) model
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.019, ANOVA; ANOVA with treatment and race (Japanese versus non-Japanese) as factors adjusted for clustered observations (from each of the participant's eyes); Mean Difference = -0.25, 95% CI 2-sided [-0.46 to -0.04] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Change in Vitreous Haze (VH) Grade in Each Eye From Best State Achieved Prior to Week 6 to the Final/Early Termination Visit
Description: Vitreous haze was measured using dilated indirect ophthalmoscopy (DIO) and assessed by the Investigator according to National Eye Institute (NEI) and SUN criteria:
  Grade 0: No evident vitreous haze;
  Grade 0.5+: Slight blurring of the optic disc margin because of the haze; normal striations and reflex of the nerve fiber layer cannot be visualized;
  Grade 1+: Permits a better definition of both the optic nerve head and the retinal vessels (compared to higher grades);
  Grade 2+: Permits better visualization of the retinal vessels (compared to higher grades);
  Grade 3+: Permits the observer to see the optic nerve head, but the borders are quite blurry;
  Grade 4+: Optic nerve head is obscured.
Time Frame: From Baseline to Week 6 and Final/Early Termination Visit (up to 80 weeks)
Population: Intent-to-treat population with values at both time points; last observation carried forward (LOCF) imputation was used; participants with no values after Week 6 were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 103 | 101 | 111 | 109
units on a scale
  Left Eye | 0.33 (0.666) | 0.11 (0.559) | 0.34 (0.675) | 0.11 (0.547)
  Right Eye | 0.45 (0.781) | 0.13 (0.648) | 0.49 (0.815) | 0.16 (0.648)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with treatment as factor adjusted for clustered observations; Mean Difference = -0.27, 95% CI 2-sided [-0.43 to -0.11] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with treatment and race (Japanese versus non-Japanese) as factors adjusted for clustered observations; Mean Difference = -0.28, 95% CI 2-sided [-0.43 to -0.12] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change In Logarithm of the Minimum Angle of Resolution (LogMAR) Best Corrected Visual Acuity (BCVA) In Each Eye From Best State Achieved Prior to Week 6 to the Final/Early Termination Visit
Description: Using corrective lenses based on that visit's refraction testing, participant's best corrected visual acuity was measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart.
Time Frame: From Baseline to Week 6 and Final/Early Termination Visit (up to 80 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 103 | 101 | 111 | 109
logMAR
  Left Eye | 0.12 (0.169) | 0.07 (0.160) | 0.11 (0.179) | 0.07 (0.164)
  Right Eye | 0.13 (0.320) | 0.04 (0.143) | 0.13 (0.328) | 0.05 (0.145)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.003, ANOVA; ANOVA with treatment as factor adjusted for clustered observations; Mean Difference = -0.07, 95% CI 2-sided [-0.11 to -0.02] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.008, ANOVA; ANOVA with treatment and race (Japanese versus non-Japanese) as factors adjusted for clustered observations; Mean Difference = -0.06, 95% CI 2-sided [-0.10 to -0.02] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Time to Optical Coherence Tomography (OCT) Evidence of Macular Edema in At Least 1 Eye On or After Week 6
Description: Optical coherence tomography was performed at every visit using 1 of 3 approved machines. Images were evaluated by a central reader. Macular edema was defined as cystoid macular edema.
  OCT evidence of macular edema on or after Week 6 was to be counted as an event. Dropouts due to reasons other than OCT evidence of macular edema were to be considered as censored observations at the time of dropping out.
Time Frame: From Baseline until the Final Visit (up to 80 weeks)
Population: Intent to treat population with no macular edema at Baseline
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 45 | 55 | 47 | 57
months | 6.2 [1.4 to NA] — Could not be estimated due to the low number of events | 11.1 [2.6 to 15.9] | 3.7 [1.4 to NA] — Could not be estimated due to the low number of events | 9.2 [2.7 to 15.9]
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.231, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.39 to 1.26] — The hazard ratio of adalimumab versus placebo was calculated using proportional hazards regression with treatment as factor
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.191, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.38 to 1.21] — The hazard ratio of adalimumab versus placebo was calculated using proportional hazards regression with treatment and race (Japanese versus non-Japanese) as factors

6. Secondary Outcome: Percent Change in Central Retinal Thickness in Each Eye From Best State Achieved Prior to Week 6 to the Final/Early Termination Visit
Description: Central retinal thickness was measured using optical coherence tomography and assessed by a central reader.
Time Frame: Baseline to Week 6 and Final/Early Termination Visit (up to 80 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 102 | 101 | 108 | 109
percent change
  Left eye (n=100, 100, 107, 108) | 20.2 (52.01) | 9.6 (29.76) | 19.0 (50.57) | 13.9 (53.95)
  Right eye (n=102, 101, 108, 109) | 22.0 (62.48) | 8.2 (25.78) | 21.7 (60.75) | 14.5 (57.05)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.020, ANOVA; ANOVA with treatment and OCT machine as factors adjusted for clustered observations; Mean Difference = -11.4, 95% CI 2-sided [-20.9 to -1.8] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.428, Chi-squared, Corrected; ANOVA with treatment, race (Japanese versus non-Japanese) and OCT machine as factors adjusted for clustered observations; Mean Difference = -5.1, 95% CI 2-sided [-17.7 to 7.5] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Change in Visual Functioning Questionnaire 25 (VFQ-25) Composite Score From Best State Achieved Prior to Week 6 to the Final/Early Termination Visit
Description: The National Eye Institute VFQ-25 is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning.
  The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question. The overall composite score ranges from 0 to 100, where higher scores or increases in score indicate better vision-related functioning.
Time Frame: Baseline to Week 6 and Final/Early Termination Visit (up 80 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 102 | 101 | 110 | 109
units on a scale | -5.50 (11.968) | -1.30 (10.980) | -5.34 (11.899) | -1.68 (10.924)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.010, ANOVA; ANOVA with treatment as a factor; Mean Difference = 4.20, 95% CI 2-sided [1.02 to 7.38]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.019, ANOVA; ANOVA with treatment and race (Japanese versus non-Japanese) as factors; Mean Difference = 3.67, 95% CI 2-sided [0.62 to 6.71]

8. Secondary Outcome: Change in VFQ-25 Distance Vision Subscore From Best State Achieved Prior to Week 6 to the Final/Early Termination Visit
Description: The National Eye Institute VFQ-25 is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning.
  The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question.
  The distance vision subscore is calculated from the answers to 3 distance vision-related questions and ranges from 0 to 100, where higher scores or increases in score indicate better vision-related functioning.
Time Frame: Baseline to Week 6 and Final/Early Termination Visit (up 80 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 102 | 101 | 110 | 109
units on a scale | -5.64 (14.654) | -3.77 (13.414) | -5.72 (14.531) | -4.42 (13.871)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.346, ANOVA; ANOVA with treatment as a factor; Mean Difference = 1.86, 95% CI 2-sided [-2.03 to 5.75]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.496, ANOVA; ANOVA with treatment and race (Japanese versus non-Japanese) as factors; Mean Difference = 1.31, 95% CI 2-sided [-2.47 to 5.09]

9. Secondary Outcome: Change in VFQ-25 Near Vision Subscore From Best State Achieved Prior to Week 6 to the Final/Early Termination Visit
Description: The National Eye Institute VFQ-25 is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning.
  The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question.
  The distance vision subscore is calculated from the answers to 3 near vision-related questions and ranges from 0 to 100, where higher scores or increases in score indicate better vision-related functioning.
Time Frame: Baseline to Week 6 and Final/Early Termination Visit (up 80 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 102 | 101 | 110 | 109
units on a scale | -8.09 (17.754) | -2.97 (16.784) | -7.65 (17.808) | -3.52 (16.494)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.036, ANOVA; ANOVA with treatment as a factor; Mean Difference = 5.12, 95% CI 2-sided [0.34 to 9.90]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.077, ANOVA; ANOVA with treatment and race (Japanese versus non-Japanese) as factors; Mean Difference = 4.14, 95% CI 2-sided [-0.45 to 8.72]

10. Secondary Outcome: Change in VFQ-25 Ocular Pain Subscore From Best State Achieved Prior to Week 6 to the Final/Early Termination Visit
Description: The National Eye Institute VFQ-25 is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning.
  The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question.
  The ocular pain subscore is calculated from the answers to 2 ocular pain-related questions and ranges from 0 to 100, where higher scores or increases in score indicate less pain.
Time Frame: Baseline to Week 6 and Final/Early Termination Visit (up 80 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 102 | 101 | 110 | 109
units on a scale | -12.62 (21.435) | -2.60 (15.342) | -12.39 (20.841) | -3.56 (16.056)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with treatment as a factor; Mean Difference = 10.02, 95% CI 2-sided [4.86 to 15.19]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with treatment and race (Japanese versus non-Japanese) as factors; Mean Difference = 8.83, 95% CI 2-sided [3.88 to 13.79]

ADVERSE EVENTS:
Time Frame: From the first study drug administration until 70 days following the last study drug administration or until rollover into the extension study. Median duration of treatment was 91 days in the placebo arm and 129 days in the adalimumab arm.
Arm/Group | Placebo | Adalimumab
Serious Adverse Events (participants affected / at risk) | 5/120 | 16/119
Other Adverse Events (participants affected / at risk) | 61/120 | 71/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | Adalimumab (N=119)
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 0 | 1
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0
PILONIDAL CYST (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0
TUBERCULOSIS (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 | 1
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
CARCINOID TUMOUR OF THE GASTROINTESTINAL TRACT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
DEMYELINATION (Nervous system disorders) | 0 | 1
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 1
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1
ABORTION INDUCED (Surgical and medical procedures) | 1 | 0
NEOVASCULARISATION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | Adalimumab (N=119)
CYSTOID MACULAR OEDEMA (Eye disorders) | 6 | 3
EYE PAIN (Eye disorders) | 2 | 9
UVEITIS (Eye disorders) | 8 | 12
VISION BLURRED (Eye disorders) | 2 | 8
DRY MOUTH (Gastrointestinal disorders) | 1 | 6
NAUSEA (Gastrointestinal disorders) | 7 | 6
FATIGUE (General disorders) | 7 | 12
BRONCHITIS (Infections and infestations) | 4 | 7
INFLUENZA (Infections and infestations) | 6 | 1
NASOPHARYNGITIS (Infections and infestations) | 11 | 21
URINARY TRACT INFECTION (Infections and infestations) | 0 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 | 10
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 9
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 | 7
HEADACHE (Nervous system disorders) | 16 | 13
PARAESTHESIA (Nervous system disorders) | 0 | 6
ANXIETY (Psychiatric disorders) | 0 | 6
INSOMNIA (Psychiatric disorders) | 8 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 7
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.